CLINICAL TRIAL: NCT00945763
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Adaptive Design, Single-Dose Study of Intravenous N1539 in the Treatment of Pain Secondary to Dental Impaction Surgery
Brief Title: Single Dose Study of N1539 in the Treatment of Pain Secondary to Dental Impaction Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N1539-02
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Dental Pain
Keywords: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Meloxicam; Sugars; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- N1539 15 mg (Experimental)
  Interventions: Drug: N1539
- N1539 30 mg (Experimental)
  Interventions: Drug: N1539
- N1539 60 mg (Experimental)
  Interventions: Drug: N1539
- Motrin (Active Comparator)
  Interventions: Drug: Motrin

INTERVENTIONS:
Drug: N1539 — 30 mg
  Other Names: meloxicam
  Arms: N1539 30 mg
Drug: placebo — tablets
  Other Names: sugar pill
  Arms: placebo
Drug: N1539 — 15 mg
  Other Names: meloxicam
  Arms: N1539 15 mg
Drug: N1539 — 60 mg
  Other Names: meloxicam
  Arms: N1539 60 mg
Drug: Motrin — 400 mg
  Other Names: ibuprofen
  Arms: Motrin

SUMMARY:
To evaluate the safety and efficacy of single IV doses of N1539 after dental impaction surgery.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single center study in subjects who have undergone third molar extraction surgery. Eligible subjects will have surgical removal of >2 third molars, of which at least 1 must be a complete or partial mandibular impaction. Each subject's study participation will consist of a screening visit (1-21 days prior to surgery), an inpatient evaluation period of 24 hours following dosing, and a follow-up phone call 3-5 days postdose.

ELIGIBILITY:
Inclusion Criteria:

* surgical extraction of > 2 third molars with at least 1 complete or partial mandibular bony extraction

Exclusion Criteria:

* allergic response to aspirin, NSAIDs, acetaminophen or hydrocodone
* use of aspirin or other analgesics within 48 hours prior to surgery
* current or recent history of drug or alcohol abuse
* any medication for treatment of chronic pain
* clinically significant abnormality on screening laboratory test active or recent history of peptic ulcer disease or GI bleeding
* prior abdominal surgery, except uncomplicated appendectomy
* any other surgical procedure within 30 days before administration of study drug
* pregnancy or breastfeeding
* untreated hypertension; SBP > 140 mmHg or DBP > 95 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Difference at End of Study | 0-24 hours

SECONDARY OUTCOMES:
Onset of action | 0-1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Steven Christensen, DDS, Principal Investigator — Jean Brown Research, Salt Lake City, UT 84124
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Viscusi ER, Gan TJ, Bergese S, Singla N, Mack RJ, McCallum SW, Du W, Hobson S. Intravenous meloxicam for the treatment of moderate to severe acute pain: a pooled analysis of safety and opioid-reducing effects. Reg Anesth Pain Med. 2019 Mar;44(3):360-368. doi: 10.1136/rapm-2018-100184. Epub 2019 Feb 7. PMID 30737315
- [Derived] Christensen SE, Cooper SA, Mack RJ, McCallum SW, Du W, Freyer A. A Randomized Double-Blind Controlled Trial of Intravenous Meloxicam in the Treatment of Pain Following Dental Impaction Surgery. J Clin Pharmacol. 2018 May;58(5):593-605. doi: 10.1002/jcph.1058. Epub 2018 Jan 12. PMID 29329493
- See also: Study site — http://www.jeanbrownresearch.com